CLINICAL TRIAL: NCT05926505
Title: Safety and Efficacy of Anakinra Treatment for Patients With Persistent Respiratory Symptoms Post Acute Covid and Immune System Activation: the Precision Double-blind, Randomized Clinical Trial
Brief Title: Safety and Efficacy of Anakinra Treatment for Patients With Post Acute Covid Syndrome
Acronym: PRECISION
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRECISION; 2023-000102-25 (EudraCT Number)
Record Dates: First submitted 2023-06-28; First posted 2023-07-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Post-Acute COVID-19 Syndrome; Post-Acute COVID-19; Long COVID
Keywords: COVID-19; Long COVID; Post-Acute COVID-19; Anakinra; PRECISION; NCT05926505
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo is injected subcutaneously once daily for 4 weeks.
  Interventions: Drug: Placebo
- Anakinra (Experimental): Anakinra is injected subcutaneously as 100 mg once daily for 4 weeks.
  Interventions: Drug: Anakinra 149 MG/ML Prefilled Syringe [Kineret]

INTERVENTIONS:
Drug: Placebo — Placebo is injected subcutaneously once daily for 4 weeks. After the period of 4 weeks, patients allocated to arm 1 will be shifted to subcutaneous treatment with 100mg anakinra once daily for 4 weeks.
  Arms: Placebo
Drug: Anakinra 149 MG/ML Prefilled Syringe [Kineret] — Anakinra is injected subcutaneously as 100 mg once daily for 4 weeks. After the first period the patients will be randomized 1:1 to continue receiving subcutaneous treatment with 100mg anakinra once daily for 4 weeks or placebo once daily for 4 weeks.
  Arms: Anakinra

SUMMARY:
The PRECISION is a proof-of-concept, phase II randomized clinical trial aiming to evaluate the efficacy and safety of anakinra in patients with Post-Acute COVID Syndrome (PACS) of the pro-inflammatory respiratory phenotype. Improvement is measured by a composite endpoint, namely, the "Score of PACS progression reversal"

DETAILED DESCRIPTION:
People with COVID-19 might have sustained post-infection sequelae, known as Post-Acute Covid Syndrome (PACS). A recent consensus definition by an international panel of 265 patients, clinicians, researchers, and WHO staff suggests that post-COVID-19 condition occurs in individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset, with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis. Common symptoms include fatigue, shortness of breath, and cognitive dysfunction and generally have an impact on everyday functioning.

The role of immune dysregulation in PACS is indirectly supported from the findings of the SAVE-MORE randomized clinical trial, in which patients with moderate and severe COVID-19, were 1:2 randomized to treatment with placebo or anakinra once daily for 10 days. The primary endpoint was the distribution of the frequencies of patients in the 11 points of the WHO clinical progression scale (CPS) by day 28. Patients' follow-up until day 90 showed significant reduction of the incidence of PACS; this was 24.4% among placebo-treated patients and 15.7% among patients treated with anakinra.

After the end of the SAVE-MORE trial, the understanding of the immune activation of PACS and the development of tools for the evaluation of patients have become the main aims of the Hellenic Institute for the study of sepsis (HISS) group. More precisely, patients with medical history of COVID-19 pneumonia during three separate time periods and matched comparators for age, sex, comorbidities, and state of vaccination were followed up and evaluated for PACS. Main findings can be summarized as follows:

1. For at least one year after acute COVID-19 there is considerable immune dysregulation involving both the innate and the adaptive responses.
2. Patients with PACS may be classified into four main phenotype clusters: fatigue involving 70.8%, respiratory cluster involving 33.2%, systemic symptoms involving 17.7% and other symptoms involving 26.1%.
3. The risk for progression into PACS was significantly lower among patients treated with anakinra in the acute stage (odds ratio 0.59, p: 0.017) showing a role of IL-1 for the progression into PACS.
4. Patients with fatigue bring distinct immunotype compared to the respiratory cluster.
5. IP-10 (interferon-gamma-induced protein-10) at levels more than 250 pg/ml has sensitivity 99.3%, specificity 90.9%, positive predictive value (PPV) 97.9% and negative predictive value (NPV) 97.6% for the diagnosis of the post acute COVID immune dysregulation.

PRECISION is a proof-of-concept, randomized clinical trial (RCT) aiming to evaluate the efficacy and safety of anakinra in patients with PACS in improving the clinical and immunological state over 4 to 8 weeks as measured by a composite endpoint, namely, the "Score of PACS progression reversal".

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or above 18 years
2. Male or female gender
3. In the case of women of childbearing age and men, an adequate method of contraception should be used during the study. Contraception should be maintained for at least a period of 3 months after the discontinuation of treatment. As an adequate method of contraception, it is suggested: -male or female condom with or without spermicide -contraceptive cap, a diaphragm or contraceptive sponge with a spermicide Prior to admission to the study, a pregnancy test will be performed to exclude pregnancy to women of childbearing age.
4. Written informed consent provided by the patient. For subjects without decision-making capacity, informed consent must be obtained from a legally designated representative following the national legislation in the Member State where the trial is planned.
5. History of confirmed COVID-19 infection the last 90 days or more
6. Symptoms compatible with PACS (defined as at least one positive answer to the questionnaire for restriction of daily activities) lasting for more than 2 months
7. Serum levels of IP-10 more than 250 pg/ml
8. Presence of ONE of the following two clinical conditions: Condition 1: Impaired Lung Function tests (defined as: DLCOcor <76% AND TLC and/or FVC lower than 80% of predicted) Condition 2: At least a total radiology score in HRCT more than 20 OR walking of a distance less than 500m in the 6-minute walk test

If patients meet the criteria for both Conditions 1 and 2, they will be considered for randomization and evaluation for the primary endpoint as in Condition 1.

Exclusion Criteria:

1. Age below 18 years
2. Denial for written informed consent
3. Any stage IV malignancy
4. Any primary immunodeficiency
5. Less than 1,500 neutrophils/mm3
6. Known hypersensitivity to anakinra
7. Known lung fibrosis prior to COVID-19
8. Medical history of pulmonary hypertension or chronic heart failure
9. Known chronic obstructive pulmonary disease GOLD stage 3 or 4 prior to COVID-19
10. Known active tuberculosis (under treatment) or latent tuberculosis (by positive tuberculin test)
11. Oral or IV intake of corticosteroids at a daily dose equal or greater than 0.4 mg/kg prednisone for a period greater than the last 15 days.
12. Any anti-cytokine biological treatment the last one month
13. Severe hepatic failure defined as Child-Pugh stage of 3
14. End-stage renal failure necessitating hemofiltration or peritoneal hemodialysis
15. Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study
16. Participation in any other interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Score of PACS progression reversal | Through study completion,an average of 2 years
  A positive score is defined differently for patients enrolled in the study because of Condition 1 or Condition 2. For patients enrolled in Condition 1, a positive score comprises at least two of the following: 1. At least 20% improvement of restrictive lung disease from baseline 2.No need for hospitalization οr admission to the Emergency Department 3. No increase of the degree of lung fibrosis score in lung HRCT For patients enrolled in Condition 2, a positive score comprises at least two of the following: 1. At least 20% decrease of the total score in lung HRCT OR Improved exercise capacity in the 6min walk test. 2.No need for hospitalization οr admission to the Emergency Department. 3.No increase of the degree of lung fibrosis score in lung HRCT.
  The proportion of patients achieving the above composite endpoint compared to placebo at week 4 will be the primary study endpoint.

SECONDARY OUTCOMES:
The frequency of the Score of PACS progression reversal between patients receiving 8 weeks anakinra treatment compared to patients receiving 4 weeks anakinra treatment (+4 weeks of placebo). | Through study completion,an average of 2 years
  The frequency of the Score of PACS progression reversal between patients receiving 8 weeks anakinra treatment compared to patients receiving 4 weeks anakinra treatment (+4 weeks of placebo).
Changes of concentration of cytokines produced by stimulated PBMCs at week 4 between the two arms of treatment. | Through study completion,an average of 2 years
  Changes of concentration of cytokines produced by stimulated PBMCs at week 4 between the two arms of treatment.
Change of each component of the score for the primary outcome at week 4 between the two arms of treatment. | Through study completion,an average of 2 years
  Change of each component of the score for the primary outcome at week 4 between the two arms of treatment. Post-acute COVID-19 syndrome (PACS) score. The higher the score, the worst the patients' outcome. PACS score ranges between 0-16.
At least 10% decrease of the pulmonary artery pressure at week 4 between the two arms of treatment. | Through study completion,an average of 2 years
  At least 10% decrease of the pulmonary artery pressure at week 4 between the two arms of treatment.
At least 10% increase of LV ejection fraction (if abnormal at baseline) at week 4 between the two arms of treatment. | Through study completion,an average of 2 years
  At least 10% increase of LV ejection fraction (if abnormal at baseline) at week 4 between the two arms of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarelos-Bourboulis, MD,PhD, Study Chair — Hellenic Institute for the Study of Sepsis
Locations (24):
- Out-patient long-COVID department, Jena University Hospital, Jena, Germany
- Greece (16):
  - Out-patient long-COVID department, Patras University General Hospital, Pátrai, Achaia
  - Out-patient long-COVID department III, Evangelismos Athens General Hospital, Athens, Attica
  - Out-patient long-COVID department I, Sotiria Athens Hospital of Chest Diseases, Athens, Attica
  - Out-patient long-COVID department II, Sotiria Athens Hospital of Chest Diseases, Athens, Attica
  - Out-patient long-COVID department IV, Sotiria Athens Hospital of Chest Diseases, Athens, Attica
  - Out-patient long-COVID department, Laiko General Hospital, Athens, Attica
  - 2nd Department of Propedeutic Medicine, ATTIKON University General Hospital, Chaïdári, Attica
  - 4th Department of Internal Medicine, ATTIKON University General Hospital, Chaïdári, Attica
  - Out-patient long-COVID department, Ioannina University General Hospital, Ioannina, Ioannina
  - Out-patient long-COVID department, Tzaneion Piraeus General Hospital, Piraeus, Piraeus
  - Out-patient long-COVID department, Alexandroupolis University General Hospital, Alexandroupoli
  - Out-patient long-COVID department X, Sotiria Athens Hospital of Chest Diseases, Athens
  - Out-patient long-COVID department, University Hospital of Larissa, Larissa
  - Out-patient long-COVID department II, Thriasio General Hospital of Elefsina, Magoula
  - Out-patient long-COVID department I, Thriasio General Hospital of Elefsina, Magoula
  - Out-patient long-COVID department, AHEPA Hospital of Thessaloniki, Thessaloniki
- Italy (6):
  - Infectious Diseases Clinic, Ospedale Policlinico San Martino IRCCS and Department of Health Sciences, University of Genova, Genoa, Italy, Genova
  - Department of Internal Medicine, Hospital of Jesolo, Italy, Jesolo
  - Unit of Immunology, Rheumatology, Allergy and Rare Diseases (UnIRAR), IRCCS Ospedale San Raffaele & Vita-Salute San Raffaele University, Milan, Italy, Milan
  - Infectious Diseases Clinic, University of Modena, Italy, Modena
  - Dipartimento Scienze di Laboratorio e Infettivologiche - Fondazione Policlinico Gemelli IRCCS, Roma Italy, Rome
  - ID Respiratory Unit, Spallanzani Institute of Rome, Italy, Rome
- Department of Pulmonary Medicine, Barcelona University Hospital, Barcelona, Spain